CLINICAL TRIAL: NCT03879759
Title: The Efficacy and Neurobehavioural Mechanism of N-acetyl Cysteine for Alcohol Dependence: An Exploratory Pilot Study
Brief Title: The Efficacy and Neurobehavioural Mechanism of N-acetyl Cysteine (NAC) for Alcohol Dependence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South West Sydney Local Health District (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); University of Sydney (Other)
Responsible Party: Principal Investigator, Professor Paul Haber, Clinical Director, South West Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X17-0343
Record Dates: First submitted 2019-03-10; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Study 1: NAC vs Placebo (PL) (4 weeks outpatient) Study 2: NAC vs PL (3 days inpatient) Study 2: NAC vs PL (neuromaging session before vs after treatment)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): NAC - Relapse Prevention (4 wks)
  Interventions: Drug: NAC 2400mg/day
- Arm 2 (Placebo Comparator): NAC - Relapse Prevention (4 wks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NAC 2400mg/day — 2400mg/day 2 x 600mg b.d
  Arms: Arm 1
Drug: Placebo — 4 matched placebo tablets/day
  Arms: Arm 2

SUMMARY:
The study will explore the efficacy and tolerability of a regimen of NAC (2400 mg) versus placebo for the treatment of alcohol dependence.

DETAILED DESCRIPTION:
Study 1: Relapse prevention: This is a double-blind, randomized, placebo-controlled clinical trial in which participants will receive oral NAC (2400 mg: 2x 600mg tablets twice per day) or matching placebo. Trial participants will receive either oral NAC ( dose stated above) or matching placebo for up to 4 weeks.

Study 2: Withdrawal: Trial participants will receive oral NAC (dose stated above) or matching placebo within the first 24 hours of their admission for up to 3 days.

Study 3: Participants from the relapse prevention substudy will also receive 30-minute non-invasive brain imaging session prior to and after completing the treatment regime in Study 1.

Both males and females will be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 65 meeting DSM-IV criteria for current alcohol use disorder (this is an exclusion for the healthy control sample)
* Able to understand and sign written informed consent
* Must have a stable residence and be able to identify an individual who could locate subject if needed
* Admitted for medical detoxification from alcohol (withdrawal study only)
* Blood alcohol concentration of 0.00 (if completing brain imaging session)
* Express a desire to achieve abstinence or to greatly reduce alcohol consumption (relapse prevention study only)

Exclusion Criteria:

* Clinically significant comorbidities or medical disease that might interfere with the evaluation of the study medication or present a safety concern.
* Pregnant women and women of childbearing potential who do not practice a medically acceptable form of birth control
* Women who are breastfeeding
* Dependence on any substance other than nicotine
* Court-mandated participation in alcohol treatment or pending incarceration (relapse prevention study only)
* Treatment/ingestion during the previous week of benzodiazepines or other sedative-hypnotic medications or history of recent chronic treatment with sedative-hypnotic medications (withdrawal study only)
* Dependence on any substance other than nicotine

The following exclusion criteria are only applicable to participants undergoing the brain imaging session:

* Extreme obesity
* Pregnant or have any reason to believe they are pregnant;
* Previous brain surgery;
* Ever employed as a machinist, a welder or a metal worker;
* Epilepsy
* Metal items such as pacemakers; aneurysm clips in the brain; metal dental implants; metallic fragments in the eye or anywhere else; insulin pump; metal implants; hearing aid or a prosthetic device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Study 1: Alcohol consumption | 4 weeks
  as measured by the number of heavy drinking days per week and number of drinks per drinking day
Study 1: Alcohol consumption | 4 weeks
  as measured by the abstinence rate, time to relapse and time to lapse
Study 2: Amount of Benzodiazepines administered | 3 days
  as measured by the number of benzodiazepines administered in the NAC vs placebo groups
Study 2: Amount of Benzodiazepines administered | 3 days
  as measured by Alcohol Withdrawal Scale (AWS) score
Study 2: Amount of Benzodiazepines administered | 3 days
  as measured by Visual Analogue Scale (VAS) score
Study 2: Amount of Benzodiazepines administered | 3 days
  as measured by Alcohol Urge Questionaire (AUQ) Score
Study 3: Markers of neural inflammation and responses to alcohol cue | 4 weeks
  as measured by differences in cortical levels of glutathione
Study 3: Markers of neural inflammation and responses to alcohol cue | 4 weeks
  as measured by differences in cortical levels of N-acetylaspartate
Study 3: Markers of neural inflammation and responses to alcohol cue | 4 weeks
  as measured by blood oxygen level dependent (BOLD) brain activation differences to alcohol cues (alcohol cue activation)

SECONDARY OUTCOMES:
Alcohol craving | 4 weeks
  as measured by Penn Alcohol Craving Scale (PACS) score
Mood | 4 weeks
  as measured by Depression Anxiety Stress Scale (DASS) score

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Haber, MBBS, Principal Investigator — Sydney Local Health District; Andrew Baille, PhD, Principal Investigator — Macquarie University; Kirsten Morley, PhD, Principal Investigator — University of Sydney; Warren B Logge, PhD, Principal Investigator — Sydney Local Health District
Locations (1):
- Drug Health Services, Royal Prince Alfred Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Dunbar KY, Dali G, DeMayo MM, Logge W, Hurzeler T, Kelly C, Watt J, Squeglia LM, Kirkland AE, Haber PS, Morley KC. The Effect of N-Acetylcysteine (NAC) on Neurometabolites and Cognitive Function in Adults With Alcohol Use Disorder: A Preliminary Randomized Controlled Trial. Neuropsychopharmacol Rep. 2025 Dec;45(4):e70066. doi: 10.1002/npr2.70066. PMID 41128676
- [Derived] Logge WB, Haber PS, Hurzeler TP, Towers EE, Morley KC. The effects of N-acetyl cysteine on intrinsic functional connectivity and neural alcohol cue reactivity in treatment-seeking individuals with alcohol use disorder: a preliminary study. Psychopharmacology (Berl). 2025 Jan;242(1):149-160. doi: 10.1007/s00213-024-06656-z. Epub 2024 Aug 5. PMID 39102049